CLINICAL TRIAL: NCT00002180
Title: A Phase I/II Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerance, and Pharmacokinetics, and Antiviral Activity of 9-[(R)-2-(Phosphonomethoxy)Propyl] Adenine (PMPA) in HIV-Infected Patients
Brief Title: A Study of PMPA in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 269A; GS-96-701
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-09

CONDITIONS: HIV Infections
Keywords: Placebos; Anti-HIV Agents; Adenine
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir

SUMMARY:
The purpose of this study is to see if it is safe and effective to give PMPA to HIV-infected patients. This study also examines how the body handles PMPA.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Laboratory diagnosis of HIV infection.
* CD4 cell count >= 200 cells/mm3 within 28 days prior to entry.
* Plasma HIV RNA >= 10,000 copies/ml within 28 days of entry.
* Minimum life expectancy of 12 months.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Active, serious infections (other than HIV) that require parental antibiotic therapy. Patients may be considered recovered if at least 2 weeks have elapsed following cessation of parental therapy before enrollment.
* Active clinically significant medical problems that include cardiac disease (e.g., symptoms of ischemia, congestive heart failure, or arrhythmia).
* Positive test for Hepatitis B surface antigen or Hepatitis C antibody in serum.

Patients with any of the following prior conditions are excluded:

History of malignancy other than basal cell carcinoma or cutaneous Kaposi's sarcoma.

Patients who are receiving:

* Antiretroviral therapy, including nucleoside analogs, non-nucleoside reverse transcriptase inhibitors, protease inhibitors or investigational antiretroviral agents.
* Interferon or interleukin therapy, aminoglycoside antibiotics, amphotericin B, cidofovir, diuretics, foscarnet, ganciclovir, itraconazole, fluconazole, ketoconazole (topical allowed), isoniazid, rifampin, rifabutin, clarithromycin, azithromycin, systemic chemotherapeutic agents, systemic corticosteroids, other agents with significant nephrotoxic potential, other agents that may inhibit or compete for elimination via active renal tubular secretion (probenecid) and other investigational agents.

Within 2 weeks prior to entry:

* Antiretroviral therapy, including nucleoside analogs, non-nucleoside reverse transcriptase inhibitors, protease inhibitors or investigational antiretroviral agents.
* Interferon or interleukin therapy, aminoglycoside antibiotics, amphotericin B, cidofovir, diuretics, foscarnet, ganciclovir, itraconazole, fluconazole, ketoconazole (topical allowed), isoniazid, rifampin, rifabutin, clarithromycin, azithromycin, systemic chemotherapeutic agents, systemic corticosteroids, other agents with significant nephrotoxic potential, other agents that may inhibit or compete for elimination via active renal tubular secretion (probenecid) and other investigational agents.

Active drug or alcohol abuse as demonstrated by a positive screening test for drugs of abuse (except marijuana or drugs used for medical indications), or substance abuse considered sufficient to hinder patient compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - San Francisco Gen Hosp / AIDS Program, San Francisco, California
  - Johns Hopkins Univ, Baltimore, Maryland